CLINICAL TRIAL: NCT06915350
Title: The Role of Maspin (Mammary Serine Protease Inhibitor) in Colorectal Carcinoma, an Immunohistochemical Study
Brief Title: The Role of Maspin in Colorectal Carcinoma, an Immunohistochemical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Salama Salah, Demonstrator, Assiut University
Other Study IDs: Maspin in colorectal carcinoma
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Maspin in Colorectal Carcinoma
MeSH Terms: interventions — SERPIN-B5

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: maspin ( mammary serine protease inhibitor) — Maspin is an immunohistochemical marker to detect the prognosis of colorectal carcinoma

SUMMARY:
Colorectal carcinoma (CRC) is a common cancer that arises from genetic and epigenetic changes in colon stem cells. The protein maspin acts as a tumor suppressor, influencing cell adhesion, motility, apoptosis, and angiogenesis. Its role varies by localization within cells; cytoplasmic maspin is associated with low metastatic risk, while nuclear maspin is linked to early recurrence in advanced CRC. Maspin's function can be either tumor-suppressive or oncogenic, depending on its expression and methylation status. Further research is needed to fully understand its prognostic significance in CRC.

DETAILED DESCRIPTION:
Colorectal carcinoma (CRC) ranks as the third most common cancer worldwide, significantly contributing to cancer-related deaths and increasingly affecting younger populations .CRC develops when stem cells present at the base of the colon crypts undergo genetic and epigenetic modifications which affect oncogenes and tumour suppressor genes, leading to the transformation of normal stem cells to cancerous stem cells .Tumor suppressor genes( TSGs) : are genes involved in DNA damage repair, inhibition of cell division, induction of apoptosis, and suppression of metastasis . Maspin(mammary serine protease inhibitor) is a protease inhibitor of the serpin family, known to have tumor suppressor activity .maspin was called a multifaced protein, because it interacts with diverse groups of intercellular and extracellular proteins, and regulates cell adhesion, motility, apoptosis, and angiogenesis.Maspin expression has been demonstrated in multiple tissues including epithelium of the breast, prostate. Depending on the cell type, maspin also demonstrates a broad localization pattern. In mammary epithelial cells, maspin localizes primarily to the cytoplasm, but can also localize to the nucleus (in myoepithelial cells), secretory vesicles, and the cell surface. The localization of maspin appears important to its function(s) since in some tissues, aberrant maspin localization can be indicative of a neoplastic lesion. demonstrated that the cytoplasmic localization of maspin in ovarian carcinoma coincided with a poor prognosis, whereas nuclear maspin localization in these cancers was indicative of a more benign lesion, suggesting an important tumor-suppressive r role for nuclear maspin. Maspin has two opposing roles in cancer, it acts as a tumor suppressor that is down-regulated in gastric, breast versus an oncogenic role as it is over-expressed in gall bladder carcinoma.

Its role as tumor suppressor gene occurs through promoter hypomethylation and histone acetylation. On the contrary, maspin promoter methylation is associated with maspin tumor suppressor gene silencing and oncogenic potentiation. To our knowledge,few studies assesed the prognostic role of maspin in colorectal carinoma . Investigators reported that the prognostic role of maspin depend on it's subcellular localization as the cytoplasmic maspin positivity is considered as an indicator of low metastatic risk and late recurrence but nuclear positivity is correlated with early recurrence after surgery, especially for advanced stage carcinomas. study will include 50 formalin-fixed parrafin embedded blocks of Colorectal carcinoma cases . Colectomy specimens will be obtained from the archive of the Surgical Pathology Laboratory Assiut University Hospital, Faculty of Medicine. The cliniopathological features will be obtained from the hospital medical records, including patient age, gender, tumor site, tumor size . Representative hematoxylin and eosin-stained slides of tumor will be examined for each specimen for identification of the following features: histologic type and grade according to WHO( World Health Organization) classification of colon and rectal tumors, 5th edition, 2019) , lympho-vasular(LVI) and perineural invasion (PNI),depth of tumor invasion, lymph node metastasis, pathologic stage (according to TNM classification of the American Joint Committee on Cancer (AJCC) 8th edition. Immunohistochemical staining:Tissue sections of 4 µm thickness of formalin-fixed paraffin-embedded specimens will be taken from tissue blocks. Sections will be deparaffinized in xylene and rehydrated in a descending graded ethanol series. The endogenous peroxidase will be blocked with 6% hydrogen peroxide. For epitope retrieval, sections will be microwaved in citrate buffer, pH 6. Then sections will be incubated with the primary antibodies (Maspin) Then the Secondary staining kits were used according to the manufacturers instructions

ELIGIBILITY:
Inclusion Criteria:

* all patients with different stages of colorectal carcinoma with available paraffin blocks and clinical data .

Exclusion Criteria:

* all cases not fulfill the inclusion criteria .

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases with different stages of colorectal adenocarcinoma with available paraffin blocks and clinical data
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
In our study we will assess the subcellular ( cytoplasmic or nuclear)expression of maspin in colorectal adenocarcinoma cases and correlate it with the prognosis | Baseline
  For the immunostains, the subcellular localization is indicated to be quantified based on the intensity, percentage and localization in the tumor cells Using a cut-off point, cases can be grouped in: negative cases, carcinomas with cytoplasm predominance (cytoplasmic high and nuclear low), nuclear expression (cytoplasmic low and nuclear high), respectively with mixed expression (dual positivity, with high cytoplasm and high nuclear intensity) and correlate this expressions with prognosis , cases with cytoplasmic predominance mean good prognosis , and cases with nuclear predominance mean poor prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Mahmoud, Assistant professor, Study Director

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menbari Oskouie I, Alemi H, Khavandgar N, Mardani-Fard HA, AleTaha A, Mousavian AH, Rahimi A, Abdollahi M, Soltani A, Kasaeian A, Sorouri M. Global Research Trends on Colorectal Cancer (2014-2023): A Scientometric and Visualized Study. Arch Iran Med. 2024 Oct 1;27(10):563-572. doi: 10.34172/aim.31944. Epub 2024 Oct 1. PMID 39492563
- [Background] Smulders-Srinivasan TK, Jenkinson SE, Brown LJ, Lenis VP, Bass R. PDIA6 and Maspin in Prostate Cancer. Anticancer Res. 2023 Dec;43(12):5331-5340. doi: 10.21873/anticanres.16736. PMID 38030170
- [Background] Shankar E, Pandey M, Verma S, Abbas A, Candamo M, Kanwal R, Shukla S, MacLennan GT, Gupta S. Role of class I histone deacetylases in the regulation of maspin expression in prostate cancer. Mol Carcinog. 2020 Aug;59(8):955-966. doi: 10.1002/mc.23214. Epub 2020 May 11. PMID 32391971
- [Background] Elkady N, Elgendy W, Badr MT, Aiad H, Samara M, Badr NM. Evaluation of the diagnostic utility of NCOA3, Maspin and VHL protein expression in pancreatic ductal adenocarcinoma: An immunohistochemical study. Ann Diagn Pathol. 2024 Dec;73:152356. doi: 10.1016/j.anndiagpath.2024.152356. Epub 2024 Jun 18. PMID 38901088
- [Background] Tang S, Lian X, Jiang J, Cheng H, Guo J, Huang C, Meng H, Li X. Tumor Suppressive Maspin-Sensitized Prostate Cancer to Drug Treatment Through Negative Regulating Androgen Receptor Expression. Front Cell Dev Biol. 2020 Oct 26;8:573820. doi: 10.3389/fcell.2020.573820. eCollection 2020. PMID 33195208
- [Background] Sakabe T, Wakahara M, Shiota G, Umekita Y. Role of cytoplasmic localization of maspin in promoting cell invasion in breast cancer with aggressive phenotype. Sci Rep. 2021 May 31;11(1):11321. doi: 10.1038/s41598-021-90887-z. PMID 34059749
- [Background] Wang N, Chang LL. Maspin suppresses cell invasion and migration in gastric cancer through inhibiting EMT and angiogenesis via ITGB1/FAK pathway. Hum Cell. 2020 Jul;33(3):663-675. doi: 10.1007/s13577-020-00345-7. Epub 2020 May 14. PMID 32409959
- [Background] Shi S, Zhang ZG, Sang YZ, Sun J, Ma HY. A meta- and bioinformatics analysis of maspin expression levels influencing the prognosis of patients with breast cancer. Oncol Lett. 2024 Feb 23;27(4):173. doi: 10.3892/ol.2024.14306. eCollection 2024 Apr. PMID 38464336
- [Background] Baghel K, Kazmi HR, Chandra A, Raj S, Srivastava RN. Significance of methylation status of MASPIN gene and its protein expression in prognosis of gallbladder cancer. Asia Pac J Clin Oncol. 2019 Oct;15(5):e120-e125. doi: 10.1111/ajco.13129. Epub 2019 Feb 10. PMID 30740890
- [Background] Marioni G, Ottaviano G, Lovato A, Franz L, Bandolin L, Contro G, Giacomelli L, Alessandrini L, Stramare R, de Filippis C, Blandamura S. Expression of maspin tumor suppressor and mTOR in laryngeal carcinoma. Am J Otolaryngol. 2020 Jan-Feb;41(1):102322. doi: 10.1016/j.amjoto.2019.102322. Epub 2019 Oct 23. PMID 31732312